CLINICAL TRIAL: NCT05107063
Title: A Multi-center, Prospective Observational Study to Investigate the Effectiveness of Pravastatin on Renal Function in Korean Dyslipidemic Patients With Type 2 Diabetes
Brief Title: An Observational Study Investigating the Effectiveness of Pravastatin on Renal Function in Korean Dyslipidemic Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MVT-OS-15-01
Record Dates: First submitted 2021-10-27; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Dyslipidemia; Type II Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2 | interventions — Pravastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyslipidemic participants with Type 2 diabetes: Dyslipidemic participants with Type 2 diabetes who received a routine initiation dose of pravastatin 10 mg, 20 mg or 40 mg single dose once daily and maintained a low cholesterol diet throughout the study period.
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Routine initiation dose was 10 mg, 20 mg or 40 mg single dose once daily. Depending on patient response, dose could have been increased up to 40 mg. Maintenance dose was 10-40 mg once daily.

SUMMARY:
This study investigated the effectiveness of pravastatin on renal function in Korean dyslipidemic patients with Type 2 diabetes.

DETAILED DESCRIPTION:
This survey study investigated the effect of routine initiation single dose of pravastatin (10 mg, 20 mg, or 40 mg) on renal function in Korean dyslipidemic patients with Type 2 diabetes. The study also examined the effect of pravastatin on lipid profiles, glucose metabolism, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 diabetes (currently using an antidiabetic drug or satisfying diagnostic criteria of diabetes as defined by American Diabetes Association)
* Participants with dyslipidemia (currently using an antidyslipidemic drug or satisfying the Health Insurance Review & Assessment Service insurance coverage treatment criteria*) for whom drug treatment with pravastatin is confirmed
* Participants determined to be eligible as subjects at the discretion of the investigator
* Participants who voluntarily provided written consent using the Informed Consent Form on Use of Information

Exclusion Criteria:

* Participants who had administered pravastatin prior to study participation
* Participants with hypersensitivity to the investigational product or its history
* Participants with an active liver disease or persistent elevation of transaminase with an unknown cause
* Pregnant woman or women with childbearing potential, breastfeeding mothers
* Children
* Participants with severe hepatic or renal insufficiency
* Participants with myopathy
* Participants with cholestasis
* Participants with hypercholesterolemia due to hyperalphalipoproteinemia accompanied by HDL cholesterol elevation
* Participants with a genetic problem such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included Korean dyslipidemic participants with Type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 2972 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Percentage Change Rate From Baseline in the Modification of Diet in Renal Disease(MDRD) Estimated Glomerular Filtration Rate (eGFR) at Week 24 After Routine Care of Pravastatin Administration | Week 24 post-dose
  The following formula was used to calculate MDRD eGFR:
  MDRD eGFR (mL/min/1.73 m^2) = 186 x (serum creatinine) -1.154 x (age)-0.203 x (0.742 if female)

SECONDARY OUTCOMES:
Change from Baseline in Modification of Diet in Renal Disease (MDRD) Estimated Glomerular Filtration Rate (eGFR) at Week 24 After Routine Care of Pravastatin Administration | Week 24 post-dose
  The following formula was used to calculate MDRD eGFR:
  MDRD eGFR (mL/min/1.73 m^2) = 186 x (serum creatinine)^-1.154 x (age)^-0.203 x (0.742 if female)
Percentage Change Rate from Baseline in Modification of Diet in Renal Disease (MDRD) Estimated Glomerular Filtration Rate (eGFR) at Week 12 and Week 48 After Routine Care of Pravastatin Administration | Week 12 and Week 48 post-dose
  The following formula was used to calculate MDRD eGFR:
  MDRD eGFR (mL/min/1.73 m^2) = 186 x (serum creatinine)^-1.154 x (age)^-0.203 x (0.742 if female)
Change from Baseline in Modification of Diet in Renal Disease (MDRD) Estimated Glomerular Filtration Rate (eGFR) at Week 12 and Week 48 after Routine Care of Pravastatin Administration | Week 12 and Week 48 post-dose
  The following formula was used to calculate MDRD eGFR:
  MDRD eGFR (mL/min/1.73 m^2) = 186 x (serum creatinine)^-1.154 x (age)^-0.203 x (0.742 if female)
Percentage Change Rate from Baseline in Estimated Glomerular Filtration Rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration(CKD-EPI) Formula at Week 12, Week 24, and Week 48 After Routine Care of Pravastatin Administration | Week 12, Week 24, and Week 48 post-dose
  The following formula was used to calculate CKD-EPI eGFR:
  CKD-EPI eGFR (mL/min/1.73 m^2) = 141 × min (serum creatinine/k, 1)^α × max (serum creatinine/k, 1)^-1.209 × 0.993^(age) × 1.018 (if female), where k is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates minimum serum creatinine/k or 1, and max indicates maximum serum creatinine/k or 1.
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) using the Chronic Kidney Disease Epidemiology Collaboration(CKD-EPI) Formula at Week 12, Week 24, and Week 48 After Routine Care of Pravastatin Administration | Week 12, Week 24, and Week 48 post-dose
  The following formula was used to calculate CKD-EPI eGFR:
  CKD-EPI eGFR (mL/min/1.73 m^2) = 141 × min (serum creatinine/k, 1)^α × max (serum creatinine/k, 1)^-1.209 × 0.993^(age) × 1.018 (if female), where k is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates minimum serum creatinine/k or 1, and max indicates maximum serum creatinine/k or 1.
Percentage Change Rate from Baseline in Total Cholesterol, Low Density Lipoprotein Cholesterol, High Density Lipoprotein-Cholesterol, Triglycerides, Fasting Plasma Glucose at Week 12, Week 24, and Week 48 After Routine Care of Pravastatin Administration | Week 12, Week 24, and Week 48 post-dose
  Blood plasma samples will be collected to assess lipids (total cholesterol [mg/dL], low density lipoprotein cholesterol (LDL-C) [mg/dL], high density lipoprotein-cholesterol (HDL-C) [mg/dL], triglyceride [mg/dL], and fasting plasma glucose [mg/dL]).
Change from Baseline in Total Cholesterol, Low Density Lipoprotein Cholesterol, High Density Lipoprotein-Cholesterol, Triglycerides, Fasting Plasma Glucose at Week 12, Week 24, and Week 48 After Routine Care of Pravastatin Administration | Week 12, Week 24, and Week 48 post-dose
  Blood plasma samples will be collected to assess lipids (total cholesterol [mg/dL], low density lipoprotein cholesterol (LDL-C) [mg/dL], high density lipoprotein-cholesterol (HDL-C) [mg/dL], triglyceride [mg/dL], and fasting plasma glucose [mg/dL]).
Percentage Change Rate from Baseline in Hemoglobin A1c (HbA1c) at Week 12, Week 24 and Week 48 After Routine Care of Pravastatin Administration | Week 12, Week 24, and Week 48 post-dose
  Blood plasma samples will be collected to assess hemoglobin A1c (HbA1c) (%)levels.
Change from Baseline in Hemoglobin A1c (HbA1c) at Week 12, Week 24 and Week 48 After Routine Care of Pravastatin Administration | Week 12, Week 24, and Week 48 post-dose
  Blood plasma samples will be collected to assess hemoglobin A1c (HbA1c) (%)levels.
Number of Participants With Treatment-emergent Adverse Events After Routine Care of Prevastatin Administration | Week 48 post-dose
  Treatment-emergent adverse event (TEAE) is defined as an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (47):
- South Korea (47):
  - Korea University Ansan Hospital, Ansan
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Yeongnam University Medical Center, Busan
  - Inje University Busan Paik Hospital - Site 23, Busan
  - Inje University Busan Paik Hospital - Site 26, Busan
  - Bong Seng Memorial Hospital, Busan
  - Pusan National University Hospital - Site 43, Busan
  - Pusan National University Hospital - Site 49, Busan
  - Kosin University Gospel Hospital, Busan
  - Changwon Fatima Hospital, Changwon
  - Soon Chun Hyang University Cheonan Hospital, Cheonan
  - Daegu Catholic University Medical Center, Daegu
  - Eulji University DaeJeon Medical Center, Daejeon
  - Konyang University Hospital, Daejeon
  - GangNeung Asan Hospital, Gangneung
  - Dongguk University Ilsan Hospital, Goyang
  - Inje University Ilsan Paik Hospital, Goyang
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Myongji Hospital, Goyang
  - Chosun University Hospital, Gwangju
  - Gwangju Veterans Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Bundang CHA General Hospital, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - HANIL General Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Eulji University Medical Center - Site 20, Seoul
  - Eulji University Medical Center - Site 52, Seoul
  - Seoul Medical Center, Seoul
  - The Catholic University of Korea, St. Paul's Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Soon Chun Hyang University Seoul Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - VHS Medical Center, Seoul
  - Yonsei University Health System, Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang Univerisity Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - St. Carollo General Hospital, Suncheon
  - The Catholic University of Korea, St. Vincent's Hospital - Site 45, Suwon
  - The Catholic University of Korea, St. Vincent's Hospital - Site 50, Suwon
  - Ajou University Hospital - Site 04, Suwon
  - Ajou University Hospital - Site 05, Suwon
  - Dongkang Medical Center, Ulsan
  - Yonsei University, Wonju Severance Christian Hospital - Site 10, Wŏnju
  - Yonsei University, Wonju Severance Christian Hospital - Site 15, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Hur KY, Lee YH, Kim JT, Lee YK, Baek KH, Choi EJ, Hwang WM, Bang KT, Lim JS, Chung YJ, Jo SR, Oh JS, Lee SH, Ko SH, Choi SH. Effect of Pravastatin on Kidney Function in Patients with Dyslipidemia and Type 2 Diabetes Mellitus: A Multicenter Prospective Observational Study. Adv Ther. 2024 Aug;41(8):3119-3137. doi: 10.1007/s12325-024-02862-5. Epub 2024 Jun 16. PMID 38880822